CLINICAL TRIAL: NCT05377307
Title: Long-term Follow-up Study to Evaluate the Safety and Efficacy in Patients Who Have Ever Received Lentiviral-based Gene-edited Immune Cell Therapy
Brief Title: Long-term Follow-up Study of Lentiviral-based Gene-edited Immune Cell Therapy
Status: Recruiting | Type: Observational
Sponsor: Pell Bio-Med Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PLLV-LTFU-401
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Large B-cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Follicular Lymphoma Grade 3A; Follicular Lymphoma Grade 3B
Keywords: DLBCL(Diffuse Large B Cell Lymphoma); PMLBCL(Primary Mediastinal Large B Cell Lymphoma); FL(Follicular Lymphoma)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: After completion or early withdraw from the treatment protocol, patients will be enrolled into this long-term follow-up study. If patients do not enter this study right after leaving the treatment protocol, they may have the option to enter this study at any time within 15 years after the last lentiviral-based gene-edited immune cell infusion.
  Interventions: Genetic: Pell's lentiviral-based gene-edited immune cell therapy
- Group B: Some patients may require joining other Pell's gene-edited immune cell therapy study during participating in this long-term follow-up study. For such case, the patient could be enrolled into the new treatment protocol. Meanwhile, the patient can be remaining in this long-term follow-up protocol as an inactive participant.
  Interventions: Genetic: Pell's lentiviral-based gene-edited immune cell therapy

INTERVENTIONS:
Genetic: Pell's lentiviral-based gene-edited immune cell therapy — No study drug or other planned treatment will be administered. Subjects who previously received Pell's lentiviral-based gene-edited immune cell therapy will be evaluated the safety and efficacy.

SUMMARY:
According to health authorities guidances (FDA 2006, EMA(European Medicines Agency) 2009) for gene therapy clinical trials, observing subjects for delayed adverse events for 15 years is recommended. This purpose of this long-term follow-up study is to evaluate the safety and efficacy in patients who have ever received lentiviral-based gene-edited immune cells which are manufactured by Pell Bio-Med Technology Co. Ltd.

DETAILED DESCRIPTION:
After completion or early withdraw from the other treatment protocol, patients should be enrolled into this long-term follow-up study. If patients do not enter this study right after leaving the treatment protocol, they may have the option to enter this long-term follow-up study at any time within 15 years after the last lentiviral-based gene-edited immune cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have ever received Pell's lentiviral-based gene-edited immune cell as monotherapy or as combination therapy in clinical trials.
2. The last lentiviral-based gene-edited immune cell infusion within 15 years.
3. Patient/patient's parent/legal guardian is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

There are no specific exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes all patients who have ever received Pell's lentiviral-based gene-edited immune cell therapy.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2036-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
To assess delayed adverse events which are suspected related to previous gene-edited immune cell therapy | 15 years
  • Proportion of patients with any events of the following items which are suspected related to previous gene-edited immune cell therapy.
  1. New malignancies
  2. New incidence or exacerbation of a pre-existing neurologic disorder
  3. New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder
  4. New incidence of a hematologic disorder, including hypogammaglobulinemia
  5. New incidence of infection (potentially product-related)
  6. Other than the above adverse events, which are suspected related to gene-edited immune cell therapy judged by the investigator

SECONDARY OUTCOMES:
Monitor for Replication Competent of Lentivirus (RCL) | 15 years
  Proportion of patients with detectable RCL in peripheral blood by VSV-G(Vesicular stomatitis virus G) qPCR
Monitor the persistence of gene-edited immune cells in peripheral blood(By qPCR) | 15 years
  Proportion of patients with detectable transgene level in peripheral blood by qPCR
Monitor the persistence of gene-edited immune cells in peripheral blood(By Flowcytometry) | 5 years
  Persistence of gene-edited immune cells in peripheral blood using flow cytometry
To assess the long-term efficacy of gene-edited immune cells | 15 years
  1. Proportion of patients with relapse or progress among patients who didn't progress or relapse at study entry/reentry
  2. Incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Lung Lin, MD, Study Chair — Pell Bio-Med Technology Co., Ltd.
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Veterans General Hospital, Taipei, Taiwan
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No